CLINICAL TRIAL: NCT06892756
Title: Open-label, Non-randomised, Single-dose, One Sequence, Two-period, Cross-over Study to Investigate the Effect of Inhibition of P-glycoprotein and Breast Cancer Resistance Protein Transporters by Cyclosporine on the Pharmacokinetics of CHF6001 in Healthy Volunteers
Brief Title: Effect of Cyclosporine Drug Interaction on the Absorption, Metabolism and Elimination of CHF6001 in Healthy Volunteers. Drug-Drug Interaction 2 (DDI2) Study
Acronym: DDI2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLI-06001AA1-06; 2024-516475-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-05; First posted 2025-03-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: CHF6001; pharmacokinetics; healthy volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF6001 alone (Treatment Period 1) (Experimental): CHF6001 DPI (dry powder inhaler) followed by a 14 to 17-day wash-out period before Period 2
  Interventions: Drug: CHF6001 dry powder inhaler (DPI)
- CHF6001 after Cyclosporine (Treatment Period 2) (Experimental): Cyclosporine plus CHF6001
  Interventions: Drug: Cyclosporine; Drug: CHF6001 DPI

INTERVENTIONS:
Drug: CHF6001 dry powder inhaler (DPI) — CHF6001 DPI single dose administration followed by a 14 to 17-day wash-out period before Treatment Period 2
  Arms: CHF6001 alone (Treatment Period 1)
Drug: Cyclosporine — Oral cyclosporine single dose administration
  Arms: CHF6001 after Cyclosporine (Treatment Period 2)
Drug: CHF6001 DPI — CHF6001 DPI single dose administration after oral cyclosporine single dose administration
  Arms: CHF6001 after Cyclosporine (Treatment Period 2)

SUMMARY:
The main goal of this pharmacokinetic study in healthy volunteers is to evaluate the potential effect of cyclosporine (probe inhibitor of P glycoprotein [P-gp] and breast cancer resistance protein [BCRP] transporters) on CHF6001 (Tanimilast) systemic exposure following single dose administration, by comparing the area under the curve (AUC) from time 0 to the last quantifiable concentration (AUC0 t) and the maximum plasma concentration (Cmax) of CHF6001 with and without cyclosporine. Participants will receive CHF6001 alone in Treatment Period 1, then CHF6001 after oral cyclosporine in Treatment Period 2, in order to evaluate the cyclosporine drug interaction on CHF6001 systemic exposure. The two treatment periods will be separated by a wash out period of 14 to 17 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study related procedures;
2. Healthy male and female subjects aged 18 55 years inclusive;
3. Ability to understand the study procedures, the risks involved and ability to be trained to use the inhalers correctly and to generate sufficient peak inspiratory flow;
4. Body mass index between 18.0 and 30.0 kg/m2 extremes inclusive;
5. Non- or ex smokers who smoked <5 pack years;
6. Good physical and mental status determined based on the medical history and a general clinical examination, at the Screening Visit and prior to the first dosing;
7. Vital signs within normal limits at the Screening Visit;
8. A 12-lead digitalised electrocardiogram (12-lead ECG) in triplicate considered as normal at the Screening Visit;)
9. Pulmonary function test within normal limits at the Screening Visit;
10. Males fulfilling one of the following criteria:

    1. Males with pregnant or non-pregnant women of childbearing potential (WOCBP) partners: They must be willing to use male condom from the signature of the informed consent and until the Follow up Call; or
    2. Non fertile male subjects: Contraception is not required in this case; or
    3. Males with women of non childbearing potential (WONCBP) partners: Contraception is not required in this case;
11. Females fulfilling one of the following criteria:

    1. WONCBP defined as physiologically incapable of becoming pregnant. Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per Investigator's request, post menopausal status may be confirmed by follicle stimulating hormone levels;
    2. WOCBP fulfilling one of the following criteria: i. WOCBP with fertile male partners: They and/or their partner must be willing to use a highly effective birth control method preferably with low user dependency from the signature of the informed consent and until the Follow up Call; or ii. WOCBP with non fertile male partners: Contraception is not required in this case.

Exclusion Criteria:

1. Participation in another clinical study less than 8 weeks prior to the Screening Visit;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic or psychiatric disorders, gastric surgery recently or in the past, and/or impaired gastric motility that may interfere with successful completion of this protocol according to the Investigator's judgment;
3. Clinically relevant abnormal laboratory values at the Screening Visit suggesting an unknown disease and requiring further clinical investigation, or which may impact the safety of the subject or the evaluation of the results of the study according to the Investigator's judgment.
4. Abnormal liver enzymes at the Screening Visit (alanine aminotransferase or aspartate aminotransferase >1.5x upper limit of normal [ULN], bilirubin >1.5x ULN).
5. Subjects with history of breathing problems (e.g. history of asthma). Allergic asthma diagnosis in childhood (until 12 years old) is allowed;
6. Positive human immunodeficiency virus (HIV) 1 or HIV2 serology at the Screening Visit;
7. Positive results from the hepatitis serology which indicates acute or chronic hepatitis B (HB) or hepatitis C (HC) at the Screening Visit;
8. Blood donation or blood loss (≥450 mL) less than 8 weeks prior to the Screening Visit (evaluated at the Screening Visit and before the first dosing);
9. Positive urine test for cotinine at the Screening Visit and/or prior to the first dosing;
10. Documented history of alcohol abuse within 12 months prior to the Screening Visit or a positive alcohol breath test at the Screening Visit and/or prior to the first dosing;
11. Documented history of drug abuse within 12 months prior to the Screening Visit or a positive urine drug screen evaluated at the Screening Visit and/or prior to the first dosing;
12. Presence of any current infection, or previous infection that resolved less than 7 days prior to the Screening Visit and prior to the first dosing.
13. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the study;
14. Unsuitable arm veins for repeated venipuncture;
15. Heavy caffeine drinker (>5 cups or glasses of caffeinated beverages, e.g. coffee, tea, cola per day);
16. For females only: Pregnant or lactating women;
17. Subjects using e-cigarettes within 6 months before the Screening Visit;
18. Positive test for coronavirus disease 2019 (antibody test or nucleic acid test) within 14 days prior to the Screening Visit and the associated complications/symptoms, which have not resolved within 14 days prior to the Screening Visit;
19. Intake of non-permitted concomitant medications in the predefined period prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Plasma CHF6001 AUC0-t | A total of 16 blood samples will be collected at the following time points: Pre-dose, and then 15 minutes, 30 minutes, 1 hour, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours after CHF6001 administration
  PK evaluation to determine concentrations of CHF6001 when administered alone or after cyclosporine
Plasma CHF6001 Cmax | A total of 16 blood samples will be collected at the following time points: Pre-dose, and then 15 minutes, 30 minutes, 1 hour, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours after CHF6001 administration
  PK evaluation to determine concentrations of CHF6001 when administered alone or after cyclosporine

CONTACTS AND LOCATIONS:
Overall Officials: Maya Dabcheva, MD, Principal Investigator — MC Comac Medical Ltd.
Locations (1):
- Medical Centre Comac Medical Ltd, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No